CLINICAL TRIAL: NCT01043237
Title: A Single-centered Investigation Into the Frequency Domain Patterns in Vessels of Patients With Coronary Artery Disease
Brief Title: Frequency Analysis of Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 0901M57884
Record Dates: First submitted 2010-01-04; First posted 2010-01-06 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: Coronary Artery Disease
Keywords: acoustic; digital; sound; vibration; coronary; auscultation; artery; diagnosis
MeSH Terms: conditions — Coronary Artery Disease; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine if coronary artery disease can be detected using an electronic, acoustic recording instrument. The presence or absence of abnormal pathology will be confirmed by diagnostic angiography as part of the normal patient care at this institution.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-89 years old and recommended for a cardiology related angiogram within 24 hours

Exclusion Criteria:

* Any patient less than 18 years of age or greater than 89 years of age.
* Any patient with any of the following conditions: pregnant or nursing, prior myocardial infarction, left ventricular device, heart transplant, valve replacement, congestive heart failure, atrial fibrillation (non-intermittent), endocarditis or any heart viral or bacterial infection, any patient who has or requires medication or other heart rhythm altering treatment.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the University of Minnesota Medical Center (UMMC) Fairview Clinics, Physicians (UMP) or the Redwing, Minnesota clinic
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2009-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
to determine if coronary artery disease can be detected using an electronic, acoustic recording instrument | Baselin
  to determine if coronary artery disease can be detected using an electronic, acoustic recording instrument

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wilson, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center (UMMC) Fairview Clinics, Minneapolis, Minnesota, United States